CLINICAL TRIAL: NCT02141620
Title: Motivation for Cocaine and Non-Drug Reinforcers: Targeting Glutamate Homeostasis
Brief Title: n-Acetylcysteine and Cocaine
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, William Stoops, Associate Professor, University of Kentucky
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: R21DA035376 (NIH)
Record Dates: First submitted 2014-05-13; First posted 2014-05-19 (Estimated); Results first posted 2016-10-06 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine Abuse; Cocaine Dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Cocaine; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects will be maintained on oral placebo.
  Interventions: Drug: Cocaine; Drug: Placebo
- n-Acetylcysteine (Experimental): Subjects will be maintained on oral n-acetylcysteine.
  Interventions: Drug: Cocaine; Drug: n-Acetylcysteine

INTERVENTIONS:
Drug: Cocaine — The pharmacodynamic effects of cocaine will be determined during maintenance on placebo and n-acetylcysteine.
Drug: n-Acetylcysteine
  Arms: n-Acetylcysteine
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study will determine the initial efficacy, safety and tolerability of n-acetylcysteine as a pharmacotherapy for cocaine dependence. A rigorous, inpatient human laboratory study will be conducted in which the subjective, physiological and reinforcing effects of cocaine are evaluated during maintenance on placebo and n-acetylcysteine.

ELIGIBILITY:
Inclusion Criteria:

* Current cocaine use
* Current cigarette smoker

Exclusion Criteria:

* Abnormal screening outcome (e.g., ECG, blood chemistry result) that study physicians deem clinically significant
* Current or past histories of substance abuse or dependence that are deemed by the study physicians to interfere with study completion
* History of serious physical disease, current physical disease, impaired cardiovascular functioning, chronic obstructive pulmonary disease, history of seizure or current or past histories of serious psychiatric disorder that in the opinion of the study physician would interfere with study participation will be excluded from participation
* Females not currently using effective birth control
* Contraindications to cocaine or n-acetylcysteine
* History of schizophrenia in first degree relative

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-05; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kentucky Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Then n-Acetylcysteine: Subjects were maintained on placebo for 7 days, then they were crossed over to 2.4 g n-acetylcysteine daily for 7 days.
- n-Acetylcysteine Then Placebo: Subjects were maintained on 2.4 g n-acetylcysteine for 7 days, then they were crossed over to placebo daily for 7 days.
Period: Treatment Condition 1 (7 Days)
Arm/Group | Placebo Then n-Acetylcysteine | n-Acetylcysteine Then Placebo
Started | 8 | 7
Completed | 7 (7 completing subjects switched to n-acetylcysteine for Condition 2.) | 7 (7 completing subjects switched to placebo for Condition 2.)
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Condition 2 (7 Days)
Arm/Group | Placebo Then n-Acetylcysteine | n-Acetylcysteine Then Placebo
Started | 7 | 7
Completed | 7 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Completing participants.
Groups:
- All Study Participants: All subjects who completed the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (5.4)
Gender [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Times Cocaine Was Selected in the Presence of a Monetary Reward Alternative
Description: The reinforcing effects of cocaine were determined using a modified progressive ratio procedure (Stoops et al., 2010) in which subjects made 6 choices between available each available cocaine dose and money (US$0.25). Reinforcing effects are measured for each cocaine dose during both buspirone and placebo maintenance.
Time Frame: One test per cocaine dose level per intervention for each participant over his/her approximate 2 week inpatient admission.
Measure: Mean (Standard Deviation); unit: Number of Cocaine Choices
Groups:
- Placebo: Subjects were maintained on Placebo for 7 days.
- n-Acetylcysteine: Subjects were maintained on 2.4 g n-Acetylcysteine for 7 days.
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
Number of Cocaine Choices
  Placebo Cocaine | 1.0 (2.2) | 0.1 (.5)
  30 mg Cocaine | 3.4 (2.6) | 3.9 (2.4)
  60 mg Cocaine | 3.5 (2.8) | 3.9 (2.4)

2. Secondary Outcome: Peak Score on Sedative Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Sedative Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "sedative" items was summed to yield the Sedative Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: Subjects completed this measure at 15 minute intervals for 45 minutes after sampling each cocaine dose under both n-acetylcysteine and placebo maintenance conditions.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 3.8 (1.2) | 3.9 (1.4)
  30 mg Cocaine | 2.5 (.9) | 2.4 (.8)
  60 mg Cocaine | 2.6 (.92) | 2.6 (.8)

3. Secondary Outcome: Peak Score on Stimulant Subscale of the Adjective Rating Scale
Description: Subjects completed 16 items that loaded into the Stimulant Subscale of the Adjective Rating Scale. The items were rated 0-4 on a Likert-type scale and the sum for the 16 "sedative" items was summed to yield the Stimulant Subscale score. The maximum score for this scale was 64, the minimum was 0. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 6.1 (1.1) | 5.7 (1.1)
  30 mg Cocaine | 9.8 (1.4) | 9.1 (1.4)
  60 mg Cocaine | 12.2 (1.9) | 11.6 (1.5)

4. Secondary Outcome: Peak Ratings of "Active, Alert, Energetic" on the Visual Analog Scale
Description: Subjects rated their feelings of "Active, Alert, Energetic" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.4 (1.3) | .9 (.44)
  30 mg Cocaine | 14.7 (5.7) | 13.9 (4.4)
  60 mg Cocaine | 27.1 (6.6) | 20.5 (6.6)

5. Secondary Outcome: Peak Ratings of "Any Effect" on the Visual Analog Scale
Description: Subjects rated their feelings of "Any Effect" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.1 (.5) | 1.4 (.8)
  30 mg Cocaine | 19.6 (4.4) | 16.7 (4.9)
  60 mg Cocaine | 25.7 (5.8) | 28.2 (7.0)

6. Secondary Outcome: Peak Ratings of "Bad Effects" on the Visual Analog Scale
Description: Subjects rated their feelings of "Bad Effects" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.2 (.5) | 1.1 (.5)
  30 mg Cocaine | 4.2 (1.8) | 3.9 (1.7)
  60 mg Cocaine | 10.1 (4) | 7.2 (4.0)

7. Secondary Outcome: Peak Ratings of "Euphoric" on the Visual Analog Scale
Description: Subjects rated their feelings of "Euphoric" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.6 (1.5) | 1.1 (.5)
  30 mg Cocaine | 9.4 (4.3) | 3.1 (1.5)
  60 mg Cocaine | 15.1 (5.7) | 7.9 (3.7)

8. Secondary Outcome: Peak Ratings of "Good Effects" on the Visual Analog Scale
Description: Subjects rated their feelings of "Good Effects" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.1 (.4) | 1.3 (.7)
  30 mg Cocaine | 14.8 (4.4) | 16.7 (4.6)
  60 mg Cocaine | 25.3 (6.4) | 22.1 (4.6)

9. Secondary Outcome: Peak Ratings of "High" on the Visual Analog Scale
Description: Subjects rated their feelings of "High" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | .9 (.4) | 1.4 (.8)
  30 mg Cocaine | 18.2 (5.9) | 16.9 (4.4)
  60 mg Cocaine | 29.3 (6.9) | 27.1 (7.7)

10. Secondary Outcome: Peak Ratings of "Irregular/Racing Heartbeat" on the Visual Analog Scale
Description: Subjects rated their feelings of "Irregular/Racing Heartbeat" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.9 (1) | 1.1 (.53)
  30 mg Cocaine | 8.4 (3.4) | 5 (3.3)
  60 mg Cocaine | 13.6 (5.2) | 15.6 (5.6)

11. Secondary Outcome: Peak Ratings of "Like Drug" on the Visual Analog Scale
Description: Subjects rated their feelings of "Like Drug" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.4 (1.3) | 2.3 (1.3)
  30 mg Cocaine | 20.8 (5) | 19.7 (5.1)
  60 mg Cocaine | 31.7 (7.4) | 26.9 (7.1)

12. Secondary Outcome: Peak Ratings of "Nauseous" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nauseous" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | .9 (.4) | 3.9 (2.7)
  30 mg Cocaine | 2.5 (1.1) | 1.3 (.5)
  60 mg Cocaine | 8.1 (4) | 7.4 (4)

13. Secondary Outcome: Peak Ratings of "Nervous/Anxious" on the Visual Analog Scale
Description: Subjects rated their feelings of "Nervous/Anxious" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.4 (1.4) | .9 (.4)
  30 mg Cocaine | 2.3 (.9) | .9 (.4)
  60 mg Cocaine | 7.5 (3) | 9.1 (4.2)

14. Secondary Outcome: Peak Ratings of "Willing to Pay For" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Pay For" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.4 (1.8) | 3.6 (2.8)
  30 mg Cocaine | 21 (7.6) | 19.2 (6.0)
  60 mg Cocaine | 33.9 (9.5) | 31.3 (8.1)

15. Secondary Outcome: Peak Ratings of "Performance Impaired" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Impaired" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.3 (.5) | 1.4 (.6)
  30 mg Cocaine | 3.1 (1.3) | 2.9 (1.2)
  60 mg Cocaine | 3.8 (2.1) | 7 (3.6)

16. Secondary Outcome: Peak Ratings of "Performance Improved" on the Visual Analog Scale
Description: Subjects rated their feelings of "Performance Improved" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.5 (.7) | .9 (.4)
  30 mg Cocaine | 7.3 (3.4) | 6.1 (3.9)
  60 mg Cocaine | 10.1 (5.1) | 3.5 (1.6)

17. Secondary Outcome: Peak Ratings of "Restless" on the Visual Analog Scale
Description: Subjects rated their feelings of "Restless" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.0 (.42) | 1.0 (.39)
  30 mg Cocaine | 3 (1.0) | 1.1 (.4)
  60 mg Cocaine | 3.4 (1.5) | 3.2 (1.6)

18. Secondary Outcome: Peak Ratings of "Rush" on the Visual Analog Scale
Description: Subjects rated their feelings of "Rush" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.2 (.6) | .9 (.4)
  30 mg Cocaine | 12.1 (4.4) | 10.8 (4.1)
  60 mg Cocaine | 24.6 (7) | 24.8 (7.6)

19. Secondary Outcome: Peak Ratings of "Shaky/Jittery" on the Visual Analog Scale
Description: Subjects rated their feelings of "Shaky/Jittery" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.3 (1.3) | 1.3 (.7)
  30 mg Cocaine | 6.1 (2.4) | 8.1 (3.9)
  60 mg Cocaine | 14.6 (5) | 14.7 (5.5)

20. Secondary Outcome: Peak Ratings of "Sluggish/Fatigued/Lazy" on the Visual Analog Scale
Description: Subjects rated their feelings of "Sluggish/Fatigued/Lazy" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.1 (.5) | 1 (.49)
  30 mg Cocaine | 1.3 (.6) | 1.6 (.9)
  60 mg Cocaine | 4.9 (1.9) | 2.1 (1.1)

21. Secondary Outcome: Peak Ratings of "Stimulated" on the Visual Analog Scale
Description: Subjects rated their feelings of "Stimulated" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 1.1 (.4) | 1.2 (.4)
  30 mg Cocaine | 13.7 (4.2) | 7.5 (3.8)
  60 mg Cocaine | 22.1 (6.2) | 18.3 (5.6)

22. Secondary Outcome: Peak Ratings of "Willing to Take Again" on the Visual Analog Scale
Description: Subjects rated their feelings of "Willing to Take Again" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 4.2 (2.5) | 4.1 (2.4)
  30 mg Cocaine | 27.6 (7.5) | 24.9 (6.4)
  60 mg Cocaine | 35.4 (8.3) | 32.2 (8.4)

23. Secondary Outcome: Peak Ratings of "Talkative/Friendly" on the Visual Analog Scale
Description: Subjects rated their feelings of "Talkative/Friendly" on a Visual Analog Scale. This item was rated from 0 (minimum)-100 (maximum) on a Visual Analog Scale. Higher values represent greater subjective effects on this item. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 2
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
units on a scale
  Placebo Cocaine | 2.2 (1.1) | .9 (.4)
  30 mg Cocaine | 9.5 (4.4) | 11.4 (4.2)
  60 mg Cocaine | 22.3 (8.2) | 14.5 (5.3)

24. Secondary Outcome: Peak Diastolic Blood Pressure
Description: Diastolic blood pressure was measured with an automated monitor. Higher values represent greater diastolic pressure. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: This measure was completed at 15 minute intervals for 45 minutes after sampling each cocaine dose under both n-acetylcysteine and placebo maintenance conditions.
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
mm Hg
  Placebo Cocaine | 75.9 (2.2) | 74.9 (2.3)
  30 mg Cocaine | 81.1 (1.8) | 82.3 (2.4)
  60 mg Cocaine | 82.4 (3.0) | 79.9 (2.4)

25. Secondary Outcome: Peak Systolic Blood Pressure
Description: Systolic blood pressure was measured with an automated monitor. Higher values represent greater systolic pressure. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 24
Measure: Mean (Standard Error); unit: mm Hg
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
mm Hg
  Placebo Cocaine | 117.9 (2.9) | 117.2 (3.4)
  30 mg Cocaine | 128.5 (2.7) | 128.6 (3.6)
  60 mg Cocaine | 131.1 (2.7) | 127.3 (3.7)

26. Secondary Outcome: Peak Heart Rate
Description: Heart rate was measured with an automated monitor. Higher values represent greater heart rate. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 24
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
beats per minute
  Placebo Cocaine | 72.4 (1.8) | 73.6 (2.5)
  30 mg Cocaine | 82.2 (4.4) | 74.9 (2.5)
  60 mg Cocaine | 84.3 (4.3) | 85.4 (4.4)

27. Secondary Outcome: Peak Temperature
Description: Oral temperature was measured with an automated monitor. Higher values represent greater temperature. Peak scores were calculated from multiple assessments for each cocaine dose under both n-acetylcysteine and placebo conditions.
Time Frame: as for outcome 24
Measure: Mean (Standard Error); unit: degrees Fahrenheit
Arm/Group | Placebo | n-Acetylcysteine
Number analyzed (Participants) | 14 | 14
degrees Fahrenheit
  Placebo Cocaine | 98.3 (.1) | 98.3 (.1)
  30 mg Cocaine | 98.4 (.1) | 98.3 (.1)
  60 mg Cocaine | 98.3 (.1) | 98.3 (.1)

ADVERSE EVENTS:
Arm/Group | Placebo Then n-Acetylcysteine | n-Acetylcysteine Then Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 1/8 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Then n-Acetylcysteine (N=8) | n-Acetylcysteine Then Placebo (N=7)
Tooth Pain (General disorders) | 1 (1) | 0 (0) — Subject experienced tooth pain during his practice session, resulting in elevated blood pressure. This occurred prior to receiving any study doses. He was discharged from the study after his practice session.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No